CLINICAL TRIAL: NCT06487728
Title: The Validity of Urinary Titin and Skeletal Muscle Index as Predictor of Muscle Weakness in Critically Ill Patients. A Prospective Cohort Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Other Study IDs: 386/10-June 2024
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Urinary Titin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Urinary titin — Urinary titin and skeletal muscle index as predictor of muscle wasting in critically ill patient

SUMMARY:
Although skeletal muscle atrophy is common in critically ill patients, biomarkers associated with muscle atrophy have not been identified reliably. Titin is a spring-like protein found in muscles and has become a measurable biomarker for muscle breakdown and intensive care unit-acquired weakness in critically ill patients, in whom titin loss is a possible pathophysiology. The skeletal muscle index (SMI) is an alternative biomarker for muscle weakness, which is calculated by dividing the cross-sectional area (cm2) of the skeletal muscle at the level of the third lumbar vertebra by the square of the patient's height (m2) on CT The possibility of using urinary titin and skeletal muscle index for early prediction of muscle weakness in critically ill patients.

DETAILED DESCRIPTION:
All patients will be subjected to the following:

Informed consent will be obtained from patients. History taking including age, sex, comorbidities, current medications, ethnicity, reason for admission, and body mass index (BMI). General clinical examination. General laboratory investigations: (CBC, Random blood sugar, CRP, ESR).

Urinary Titin Measurement:

The first urine sample will be collected using a urethral catheter within 12 h of ICU admission and 24-hour urine samples d 24-hour urine samples on days 2, 3, 5, and 7.

Urinary titin will be measured using an ELISA kit (Maruyama et al., 2016).

Skeletal Muscle Index calculation:

This assessment calculates the skeletal muscle index (SMI) (cm2/m2) by dividing the cross-sectional area (cm2) of the skeletal muscle at the level of the third lumbar vertebra (L3) by the square of the patient's height (m2) on CT. SMI measured using CT. ( Mitobe et al. 2019).

Ultrasonographic Measurement:

Rectus femoris muscle area and diaphragm thickness will be evaluated with serial ultrasound measurements on days 1, 3, 5, and 7 of ICU admission. Recordings will be discontinued at death or ICU discharge. Cross-sectional area of the rectus femoris muscle will be evaluated at the midway between the anterior superior iliac spine and the proximal 9 end of the patella. A transducer will be placed perpendicularly to the long axis of the rectus femoris muscle with patients in the supine position under passive knee extension.

The diaphragm will be evaluated at the zone of apposition on the right chest wall. Its thickness will be measured during the end-expiration phase. Beds will be adjusted at a 30° angle. We will exclude patients whose diaphragm is unclear or difficult to measure.

Patients will be divided into three groups according to the changes in diaphragm thickness: atrophy, unchanged, and increased. A 10% change in diaphragm thickness will be regarded as the cutoff value in the three groups. Atrophy will be first classified with >10% decrease in diaphragm thickness from day 1 to the lowest value over the measurement period. Thereafter, increased thickness group will be classified when >10% increase is observed. The rest of the patients were classified into the unchanged group, as previously reported (Nakanishi et al., 2019). In the analysis, the unchanged group will be compared with atrophy and increased groups and their combination because both increased and decreased diaphragm thickness significantly influence clinical outcomes (Goligher et al., 2018). Rectus femoris cross-sectional area and diaphragm thickness will be measured thrice, and the median value was used for evaluation. All measurements will be conducted by two examiners. Intraclass and interclass correlation coefficients will be 0.99 and 0.99 for rectus femoris cross-sectional area and 0.95 and 0.95 for diaphragm thickness, respectively.

Physical Assessment and Mobilization:

When patients are awake and attentive, physical therapists will be evaluated the Medical Research Council (MRC) score and incidence of ICU-AW on days 1 and 7 of ICU admission. Intact level of consciousness and awareness will be defined by patient's response to at least three of five orders (De Jonghe et al., 2007).

ICU-AW will be defined as an MRC score of <48 on two separate occasions (Stevens et al., 2009). We will use the incidence of ICU-AW following the last measurement for comparison. 10 IMS is a measure of mobilization capabilities from 0 (lying in bed) to 10 (walking independently) (Hodgson et al., 2014). We will evaluate maximum IMS score during the study period because the maximum level of mobility is an important prognostic factor (Kim et al., 2019).

ELIGIBILITY:
Inclusion Criteria:

Consent from relatives of first degree. Consecutive adult patients who will be expected to remain in ICU for >5 days will be enrolled. Nonsurgical critically ill patients will be included because surgical insult reportedly increased urinary titin level (Tanihata et al., 2019). Age more than 18 years. Both male and female.

Exclusion Criteria:

Surgery not including percutaneous abscess drainage. Patients with expected prehospital functional status of <48 hours. Chest tube insertion, and tracheostomy in ICU. 8 Current pregnancy. Diagnosis of primary neuromuscular disease. Trauma at the measurement point.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Both sex
Study Population: Critically ill patients
Sampling Method: Non-Probability Sample
Enrollment: 161 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
The relationship between cumulative urinary titin level and rate of rectus femoris muscle atrophy on days 1 and 7 of ICU admission | At day 1 and 7 day of icu admission
  Measurement of urinary titin level and its correlation to muscle index

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Zagazig university, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF